CLINICAL TRIAL: NCT03546348
Title: Normal Value of Carrying Angle in the Elbow From Birth to Adolescents
Brief Title: Carrying Angle From Birth to Adolescents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: si684/2013
Record Dates: First submitted 2018-05-17; First posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — only measurement of the carrying angle

SUMMARY:
The carrying angle in the elbow in children is very important.Most of the results of treatment in fracture around the elbow have to measure the carrying angle.The common deformity of the elbow from cubitus varus is the change of the carrying of the elbow.There are many researches studied in normal value of the carrying angle but few had study the carrying angle from birth to adolescent.This study want to compare the carrying angle in different age and gain the knowledge of development of the carrying angle in children

DETAILED DESCRIPTION:
The study is to measure the carrying angle of the children from birth to adolescents

ELIGIBILITY:
Inclusion Criteria:

* normal children age 0 day to 16 years old
* Thai nationality

Exclusion Criteria:

* no history of fracture around the elbow or upper extremity
* no congenital anomalies or abnormal bone that interfere the upper extremity
* no genetic diseases and skeletal dysplasia
* no deformity of the elbow or upper extremity
* refuse to enrolled in the study

Ages: 1 Day to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: -all normal children who are in Bangkok are enrolled in the study .There are 17 groups start from 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15 and 16 years old including both sex.
  each group has 15 boys and 15 girls All are measured the carrying angle in both right and left elbow in full extension and supination
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
carrying angle | 1 year
  the angle between the arm and forearm in full extension and supination of the elbow

SECONDARY OUTCOMES:
age | 1 year
  age count in year

CONTACTS AND LOCATIONS:
Locations (1):
- Prof.Dr.Kamolporn Kaewpornsawan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
no sharing of the IPD data

REFERENCES:
- [Background] Baughman FA Jr, Higgins JV, Wadsworth TG, Demaray MJ. The carrying angle in sex chromosome anomalies. JAMA. 1974 Nov 4;230(5):718-20. No abstract available. PMID 4479296
- [Background] Balasubramanian P, Madhuri V, Muliyil J. Carrying angle in children: a normative study. J Pediatr Orthop B. 2006 Jan;15(1):37-40. doi: 10.1097/01202412-200601000-00008. PMID 16280718
- [Background] Beals RK. The normal carrying angle of the elbow. A radiographic study of 422 patients. Clin Orthop Relat Res. 1976 Sep;(119):194-6. PMID 954311